CLINICAL TRIAL: NCT02247596
Title: Effects of High-Dose Resveratrol on Resting Energy Expenditure and HOMA in Non-Diabetic Obese Males
Brief Title: Effects of High-Dose Resveratrol in Non-Diabetic Obese Males
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Khoo Teck Puat Hospital (Other)
Collaborators: National Medical Research Council (NMRC), Singapore (Other Government)
Responsible Party: Principal Investigator, Goh Kian Peng, PI, Khoo Teck Puat Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2009/00454
Record Dates: First submitted 2014-09-17; First posted 2014-09-25 (Estimated); Last update posted 2014-09-25 (Estimated); Status verified 2014-09

CONDITIONS: Obesity; Diabetes
Keywords: Resveratrol; obesity; insulin resistance; energy expenditure; diabetes
MeSH Terms: conditions — Obesity; Diabetes Mellitus; Insulin Resistance | interventions — Resveratrol

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Placebo (Placebo Comparator): Sugar pill 1g tds for 2 weeks
  Interventions: Drug: Placebo
- Resveratrol (Experimental): Trans-resveratrol extract from Polygonum Cuspidatum 1g three times a day for 2 weeks
  Interventions: Drug: Resveratrol

INTERVENTIONS:
Drug: Resveratrol — 1g tds 2 weeks
  Other Names: Mega Resveratrol
  Arms: Resveratrol
Drug: Placebo — Sugar pill 1g tds for 2 weeks
  Arms: Placebo

SUMMARY:
The primary aim of our study was to examine the effects of two weeks of oral resveratrol on resting energy expenditure and insulin sensitivity in non-diabetic obese male subjects. Secondary variables included plasma lipid subfraction, blood pressure and glycated hemoglobin (HbA1c).

DETAILED DESCRIPTION:
Patients were recruited between July 2009 and July 2012 from a single hospital in Singapore. Eligible patients were Chinese males, aged between 21 and 55 years old, with a body mass index (BMI) of 30 kg/m2 or more and venous glucose of <7.0 and <11.1 mmol/L at 0 and 120 minutes respectively on oral glucose tolerance testing (OGTT) following a 12-hour fast. They must be willing to abstain from embarking on an exercise regime or ingesting large quantities of resveratrol-containing foods including alcohol during the study period.

The study was a randomized, double-blind, parallel group trial consisting of a screening visit, a two-week treatment period and a post-treatment visit.

Randomization was centrally performed during treatment assignment with a 2-digit reference code placed in sealed opaque envelopes maintained by the person responsible for the preparation of the intervention drug and placebo. Trans-resveratrol extract from Polygonum Cuspidatum (Mega Resveratrol, Danbury, USA) was used in the trial. The placebo was not distinguishable by color, form, or taste from the active drug. The randomization code was unblinded only after all predefined data were recorded.

Subjects were given 1g three times a day of either resveratrol or placebo for two weeks and instructed to abstain from foods with high resveratrol content during the entire duration of the trial. Compliance was determined by pill counting at the end of the trial period. Subjects in both arms were not allowed to commence on an exercise regimen or supplements during the study period. Subjects who dropped out of the trial would not be replaced. All variables were measured at baseline and at the end of the treatment period.

RMR was measured by indirect calorimetry using a breath-by-breath metabolic gas analyser via the face-mask method.

The investigators estimated that a sample size of 18 patients per group (Total N = 36) was needed to provide 80% power and two-sided 5% to detect a difference in a Cohen's effect size of 1.0 between the two groups.

All analyses were performed using SPSS 21.0 (IBM) with statistical significance set at p < 0.05 and with the percentage change from baseline as the unit of analysis. All data were analyzed according to the intention-to-treat principle. MANOVA was performed to compare the intervention and placebo groups for the unadjusted and adjusted p-values on the study variables of interest. Normal distribution was verified with the Kolmogorov-Smirnov test and data were presented as mean ± standard deviation (SD).

ELIGIBILITY:
Inclusion Criteria:

* Ability to give informed consent
* Obese Chinese Male
* Age 21 to 55 yrs old
* No diabetes mellitus
* BMI of 30 kg/m2 or more during screening

Exclusion Criteria:

* Unwilling to abstain from ingesting large quantities of resveratrol-containing foods (eg. red wine, nuts)
* Cancer diagnosis that is currently under treatment, is clinically detectable, or that has been treated within the past 5 years
* Terminal disease or on palliative care
* Current excessive alcohol intake (>21 units per week for men; 14 units per week for women)
* Known diabetes mellitus
* Past history of unexplained hypoglycemia
* Past or current history of strokes
* History of any grape allergy
* On alternative or traditional medications
* Treated with another investigational drug within last 6 months
* Poorly controlled hypertension (SBP >/= 160 or DBP >/= 100) within last one month
* ALT and/or AST > 1.5 times above upper limit of normal within last 6 months
* GFR < 50 ml/min/1.73m2 (MDRD equation) within last 6 months
* Staff of Department of Medicine, Khoo Teck Puat Hospital

Ages: 21 Years to 55 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 36 (Actual)
Dates: Start 2009-07; Primary Completion 2012-10 (Actual); Study Completion 2012-10 (Actual)

PRIMARY OUTCOMES:
Change from baseline in Resting Energy Expenditure via indirect calorimetry at 2 weeks | 2 weeks (pre and post intervention)
  Measured in Kcal/day using a metabolic cart

SECONDARY OUTCOMES:
Change from baseline in insulin resistance via Homeostasis Model Assessment (HOMA) 2 calculator at 2 weeks | 2 weeks (pre and post intervention)
  Beta cell function, B (%),Insulin sensitivity, S (%), Insulin resistance, IR
Change from baseline in lipid subfractions at 2 weeks | 2 weeks (pre and post intervention)
  LDL, HDL and triglycerides in mmol/L
Change from baseline in Blood pressure at 2 weeks | 2 weeks (pre and post intervention)
  Systolic and diastolic blood pressure in mmHg
Change from baseline in Glycated hemoglobin at 2 weeks | 2 weeks (pre and post intervention)
  HbA1c in %

CONTACTS AND LOCATIONS:
Overall Officials: Kian Peng Goh, Principal Investigator — Khoo Teck Puat Hospital
Locations (1):
- Khoo Teck Puat Hospital, Singapore, Singapore